CLINICAL TRIAL: NCT04931576
Title: The Feasibility of no Drainage During Transoral Endoscopic Thyroidectomy Via the Vestibular Approach in Treatment of Papillary Thyroid Carcinoma
Brief Title: No Drainage During Transoral Endoscopic Thyroidectomy Vestibular Approach(TOETVA)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021-0316
Record Dates: First submitted 2021-06-14; First posted 2021-06-18 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-05

CONDITIONS: Drainage; Thyroid Cancer
Keywords: Drainage; TOETVA; Palpilary Thyroid Carcinoma; complications
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine application of drainage tube (No Intervention): After TOETVA, patients will receive one drainage tube through anterior cervical area.
- Omission of drainage tube (Experimental): After TOETVA, patients will receive complete omission of drianage tube and directly close the incision.
  Interventions: Procedure: no drainage tube applied

INTERVENTIONS:
Procedure: no drainage tube applied — No drainage tube implacement after TOETVA
  Arms: Omission of drainage tube

SUMMARY:
This study evaluates the viability and safety of no drainage tube placement during transoral endoscopic thyroidectomy vestibular approach in treatment of patients with papillary thyroid carcinoma.

DETAILED DESCRIPTION:
Transoral endoscopic thyroidectomy vestibular approach (TOETVA) is widely used due to its excellent cosmetic effect without scars on the body surface. In prevention of postoperative hemorrhage, a postoperative drainage tube is routinely placed in the surgical area. However, current opinion suggest that under the circumstance of strict and effective intraoperative hemostasis, routine application of drainage tube is unnecessary in conventional open thyroidectomy(COT). The research about drainage placement decision during endoscopic thyroidectomy is scarce currently. This study evaluates the viability and safety of no drainage tube placement during TOETVA on papillary thyroid carcinoma.

Patients allocated to the intervention group will implace no drainage tube during TOETVA and those allocated in control group will implace one drainage tube routinely.

The incidence of postoperative complications will be evaluated. The time of postoperative hospital-stay and operation time will be evaluated as well. At the same time, blood test results like WBC and CRP will be evaluated 1 day after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing thyroid surgery for the first time
2. The surgical method is TOETVA
3. There is no lateral cervical lymph node metastasis assessed before surgery
4. Fine-needle aspiration revealed palpilary thyroid carcinoma
5. It meets the surgical indications and has no obvious surgical contraindications

Exclusion Criteria:

1. previous history of thyroid surgery;
2. conventional open thyroidectomy, endoscopic thyroidectomy areola approach or axillary approach;
3. patients undergoing cervical lateral lymph node dissection;
4. past or current history of hyperthyroidism;
5. history of combined hypertension, diabetes, coagulation dysfunction, or other important organ dysfunction diseases.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
The incidence rate of hemorrhage on week 1 after surgery | 1 week
  To evaluate the incidence rate of postoperative hemorrhage (hemorrhage of surgical sites which requires reoperation)
The incidence rate of infections on week 2 after surgery | 2 week
  To evaluate the incidence rate of infections of surgical sites
The incidence rate of postoperative hematoma or seroma on week 2 after surgery | 2 week
  To evaluate the incidence rate of postoperative hematoma or seroma

SECONDARY OUTCOMES:
Pain score on day 1 after surgery | 1 day
  To evaluate the pain score via numerical rating scale on day 1 after surgery. An 11-point numeric scale (NRS 11) with 0 representing no pain and 10 representing worst pain imaginable.
Body temperature on day 1 after surgery | 1 day
  To evaluate the body temperature on day 1 after surgery.
WBC on day 1 after surgery | 1 day
  To evaluate the white blood count on day 1 after surgery.
CRP on day 1 after surgery | 1 week
  To evaluate the C-reaction protein on day 1 after surgery.
Length of post-operative hospital stay | 1 week
  To evaluate the length of post-operative hospital stay.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Schietroma M, Pessia B, Bianchi Z, De Vita F, Carlei F, Guadagni S, Amicucci G, Clementi M. Thyroid Surgery: To Drain or Not to Drain, That Is the Problem - A Randomized Clinical Trial. ORL J Otorhinolaryngol Relat Spec. 2017;79(4):202-211. doi: 10.1159/000464137. Epub 2017 Jul 15. PMID 28715809
- [Background] Soh TCF, Ong QJ, Yip HM. Complications of Neck Drains in Thyroidectomies: A Systematic Review and Meta-Analysis. Laryngoscope. 2021 Mar;131(3):690-700. doi: 10.1002/lary.29077. Epub 2020 Oct 6. PMID 33022081
- [Background] Fernandez Ranvier G, Meknat A, Guevara DE, Llorente PM, Vidal Fortuny J, Sneider M, Chen YH, Inabnet W 3rd. International Multi-institutional Experience with the Transoral Endoscopic Thyroidectomy Vestibular Approach. J Laparoendosc Adv Surg Tech A. 2020 Mar;30(3):278-283. doi: 10.1089/lap.2019.0645. Epub 2020 Jan 17. PMID 31951503